CLINICAL TRIAL: NCT02798445
Title: Clinical Trial : Terminal Axial Perforator Interruption Reflux Source (TAPIRS ) Plus Adjustable Compression System in Treatment of Venous Leg Ulcers Versus Multilayer Bandage Treatment
Brief Title: TAPIRS Technique Plus Adjustable Compression System in Treatment of Venous Leg Ulcers
Acronym: TAPIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Occidente de Kennedy (Other)
Responsible Party: Principal Investigator, ernesto nieves, vascular surgeon, md., Hospital Occidente de Kennedy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAPIRS
Record Dates: First submitted 2016-05-05; First posted 2016-06-14 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Venous Ulcer
Keywords: venous ulcer; vein; juxta cures; foam; laser
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tapirs (Experimental): this group will have surgery with endovascular laser treatment (EVLT) in the axial vein and foam sclerotherapy echo-guided in perforator veins and veins in relation with the ulcer, after the surgery the patients will have conventional wound care plus juxta cure system that give a continuous compression in the leg.
  Interventions: Other: TAPIRS
- multilayer bandage (Active Comparator): multilayer bandage and conventional wound care (grade 1A) recommendation in management of vein ulcers. gold standard
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: TAPIRS — Terminal Axial Perforator Interruption Reflux Source plus Adjustable compression system
  Arms: tapirs
Other: CONTROL — Multilayer bandages and wound care
  Arms: multilayer bandage

SUMMARY:
The aim of this study is to determine the percentage of healing of active venous ulcers following Terminal Axial Perforator Interruption Reflux Source (tapirs technique) and adjustable compression system versus a control group using the traditional multilayer bandages.

DETAILED DESCRIPTION:
Venous ulcer due to venous insufficiency causes an important morbidity to those people suffering from this condition. Most of therapies available under the obligatory health plan (POS, acronym in Spanish) to date cover the cleaning of the ulcerous lesion and its medical handling using saline solutions, topical antibiotics and elastic dressings, implying an important intake from health resources due to its chronicity and the delay in ulcers healing, which usually takes periods ranging from 12 months to several years. Therapeutic alternatives, which can guarantee optimal, fast and persistent in time healing, should be identified.

The aim of this study is to determine the percentage of healing of active venous ulcers (using a clinical, etiological, anatomic and physiopathologic classification (CEAP), C6) following Endovascular Laser Treatment (EVLT) of axial vein hypertension plus ultrasound-guided foam sclerotherapy of superficial venous reflux under knee, closing perforator veins and terminal reflux under de ulcer in patients with chronic venous ulceration (TAPIRS technique) plus compression with an adjustable compression system (juxta cures) versus a control group using the traditional multilayer bandages. The investigators expect that the minimal surgical invasive approach closing all the superficial venous reflux plus adjustable compression system will diminish the time of ulcer healing compared with standard treatment of multilayer bandage care.

ELIGIBILITY:
Inclusion Criteria:

Venous Ulcer Ulcer present for at least 4 weeks Ankle-arm index greater or equal to 0.8 mmHg

Exclusion Criteria:

Severe hepatic disease Severe cardiac disease Severe pulmonary disease Deep venous thrombosis Active participation in other clinical trials limitation in the ankle movements others limitations to move their self

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
healing rates | 12 weeks
  determine healing rates between two groups

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darvall KA, Sam RC, Bate GR, Adam DJ, Silverman SH, Bradbury AW. Photoplethysmographic venous refilling times following ultrasound guided foam sclerotherapy for symptomatic superficial venous reflux: relationship with clinical outcomes. Eur J Vasc Endovasc Surg. 2010 Aug;40(2):267-72. doi: 10.1016/j.ejvs.2010.02.025. Epub 2010 Apr 1. PMID 20362477
- [Background] Pang KH, Bate GR, Darvall KA, Adam DJ, Bradbury AW. Healing and recurrence rates following ultrasound-guided foam sclerotherapy of superficial venous reflux in patients with chronic venous ulceration. Eur J Vasc Endovasc Surg. 2010 Dec;40(6):790-5. doi: 10.1016/j.ejvs.2010.08.011. Epub 2010 Sep 27. PMID 20875753